CLINICAL TRIAL: NCT00509184
Title: Therapy of Nodal Follicular Lymphoma (Grade I/II) Clinical Stage I or II Using Involved Field Radiotherapy in Combination With Rituximab
Brief Title: Rituximab and Involved Field Radiotherapy in Early Stage Follicular Lymphoma
Acronym: MIR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Klaus Herfarth, MD (Other)
Collaborators: German Low Grade Lymphoma Study Group (Other); Roche Pharma AG (Industry)
Responsible Party: Sponsor-Investigator, Klaus Herfarth, MD, Prof. Dr. K. Herfarth, Heidelberg University
Organization: Heidelberg University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIR 2006-001212-72
Record Dates: First submitted 2007-07-30; First posted 2007-07-31 (Estimated); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Lymphoma, Malignant
Keywords: untreated
MeSH Terms: conditions — Lymphoma | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Rituximab — 375 mg/m^2, weekly (4 weeks), repeated after 4 weeks gap

SUMMARY:
Combination of involved field radiotherapy for the control of macroscopic disease and CD20 antibody Rituximab for the control of microscopic remainders in other regions in patients with early stage nodal follicular lymphoma /grade I or II). Evaluation of DFSl and toxicity.

DETAILED DESCRIPTION:
The MIR (Mabthera(R) and Involved field Radiation) study is a prospective multicenter trial combining systemic treatment with the anti CD20 antibody Rituximab (Mabthera(R)) in combination with involved field radiotherapy (30 - 40 Gy). This trial aims at testing the combination's efficacy and safety with an accrual of 85 patients.Primary endpoint of the study is progression free survival. Secondary endpoints are response rate to Rituximab, complete remission rate at week 18, relapse rate, relapse pattern, relapse free survival, overall survival, toxicity and quality of life.

More details: Witzens-Harig M, Hensel M, Unterhalt M, Herfarth K. Treatment of limited stage follicular lymphoma with Rituximab immunotherapy and involved field radiotherapy in a prospective multicenter Phase II trial-MIR trial. BMC cancer. 2011; 11: 87.

ELIGIBILITY:
Inclusion Criteria:

* verified follicular lymphoma grade 1 or 2
* only nodal involvement (incl. Waldeyer) clinical stage I or II
* largest tumor ≤ 7 cm
* adequate bone marrow reserves

Exclusion Criteria:

* ECOG >2
* Follicular lymphoma grade 3
* buky disease (>7 cm)
* involvement of the spleen
* neoplasia in PMH (except: basalioma, spinalioma)
* Immunodeficiency syndromes, viral hepatitis, connective tissue disease
* severe psychiatric disease
* pregnancy or breast feeding
* known allergies against foreign proteins

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2008-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
progression free survival | 2 years

SECONDARY OUTCOMES:
Response to Rituximab | 7 weeks
Rate of CR | 18 weeks
Toxicity (CTC Vers. 3) | 2 yrs
Relapse rate, Relapse pattern, DSF | 2 yrs
Overall survival | 2 yrs
QoL | 2 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Herfarth, MD, Principal Investigator — Heidelberg University
Locations (17):
- Germany (17):
  - Charité Campus Mitte, Berlin
  - Charité Campus Benjamin-Franklin, Berlin
  - Charité Campus Buch, Berlin
  - University of Cologne, Cologne
  - University of Dresden, Dresden
  - University of Essen, Essen
  - University of Göttingen, Göttingen
  - University of Hannover, Hanover
  - University of Heidelberg, Heidelberg
  - University of Kiel, Kiel
  - University of Mainz, Mainz
  - University of Heidelberg (Campus Mannheim), Mannheim
  - University of Marburg, Marburg
  - LMU, Munich
  - TU, Munich
  - University of Münster, Münster
  - University of Ulm, Ulm

REFERENCES:
- [Background] Witzens-Harig M, Hensel M, Unterhalt M, Herfarth K. Treatment of limited stage follicular lymphoma with Rituximab immunotherapy and involved field radiotherapy in a prospective multicenter Phase II trial-MIR trial. BMC Cancer. 2011 Feb 26;11:87. doi: 10.1186/1471-2407-11-87. PMID 21352561
- [Result] Herfarth K, Borchmann P, Schnaidt S, Hohloch K, Budach V, Engelhard M, Viardot A, Engenhart-Cabillic R, Keller U, Reinartz G, Eich HT, Witzens-Harig M, Hess CF, Dorken B, Durig J, Wiegel T, Hiddemann W, Hoster E, Pott C, Dreyling M. Rituximab With Involved Field Irradiation for Early-stage Nodal Follicular Lymphoma: Results of the MIR Study. Hemasphere. 2018 Nov 30;2(6):e160. doi: 10.1097/HS9.0000000000000160. eCollection 2018 Dec. PMID 31723798
- See also: German low grade lymphoma study group — http://www.glsg.de
- See also: German network for malignant lymphomas — http://www.lymphome.de